CLINICAL TRIAL: NCT01916837
Title: Genomic Grade Index (GGI): Feasibility in Routine Practice and Impact on Treatment Decisions in Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1668; 2009-015521-36 (EudraCT Number)
Record Dates: First submitted 2013-07-30; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Invasive Breast Cancer
Keywords: Breast cancer; Feasibility; Genomic grade index
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This study includes the collection of fresh-frozen tumor biopsies at the time of breast cancer surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm: Fresh tumor specimens were sampled prior to adding any fixative and within one hour of breast cancer surgery.
  Interventions: Other: Sampling of tumor tissue; Other: Sampling of tumor tissue after breast cancer surgery; Procedure: Sampling of tumor tissue after breast cancer surgery

INTERVENTIONS:
Other: Sampling of tumor tissue — Fresh tumor specimens were sampled prior to adding any fixative and within one hour of breast cancer surgery
Other: Sampling of tumor tissue after breast cancer surgery — Fresh tumor specimens were sampled prior to adding any fixative and within one hour of breast cancer surgery
Procedure: Sampling of tumor tissue after breast cancer surgery — Fresh tumor specimens were sampled prior to adding any fixative and within one hour of surgery

SUMMARY:
In this prospective study the investigators sought to evaluate the feasibility of using the genomic signature - Genomic Grade Index (GGI) - in routine clinical practice and its impact on treatment recommendations.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the feasibility of implementing Genomic Grade Index (GGI) in community hospitals in Belgium for breast cancer patients with node negative and 1-3 node positive early breast cancer. GGI would be considered a feasible genomic test if results were obtained in > 70% of evaluated patients.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed invasive breast cancer meeting the following criteria:

* T1, T2, or operable T3 disease
* Zero to three positive lymph nodes and no distant metastases
* Operable disease - Must have undergone breast-conserving surgery or mastectomy with either a sentinel node procedure or full axillary clearance

Exclusion Criteria:

* No other invasive cancer within the past 5 years except for adequately treated carcinoma in situ of the cervix or non melanoma skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude entering into a clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients diagnosed with early-stage invasive breast cancer and operable disease.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The success rate in obtaining the Genomic Grade Index in clinical practice | 12 months
  To evaluate the feasibility of implementing Genomic Grade Index in community hospitals in Belgium for breast cancer patients diagnosed with node negative and 1-3 node positive early-stage invasive breast cancer

SECONDARY OUTCOMES:
The impact of Genomic Grade Index results on adjuvant treatment decision | 12 months
  The secondary objective was to evaluate the impact of Genomic Grade Index on adjuvant treatment decisions for patients with early breast cancer. This was done by comparing physicians' treatment recommendations before having knowledge of the GGI test results to recommendations with a hypothetical GG-1 and GG-3 result and to the treatment ultimately administered after discussion with the patient.

OTHER OUTCOMES:
The success rate of reporting Genomic Grade Index results | 12 months
  To test the success rate of reporting GGI, a minimum sample size of 137 was calculated to have a power of 90% at a one-sided significance level of 5% using an empirical estimate of variance (null hypothesis H0: p ≤ 0.70 vs. alternative hypothesis HA: p ≥ 0.80).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

REFERENCES:
- [Derived] Metzger-Filho O, Catteau A, Michiels S, Buyse M, Ignatiadis M, Saini KS, de Azambuja E, Fasolo V, Naji S, Canon JL, Delree P, Coibion M, Cusumano P, Jossa V, Kains JP, Larsimont D, Richard V, Faverly D, Cornez N, Vuylsteke P, Vanderschueren B, Peyro-Saint-Paul H, Piccart M, Sotiriou C. Genomic Grade Index (GGI): feasibility in routine practice and impact on treatment decisions in early breast cancer. PLoS One. 2013 Aug 19;8(8):e66848. doi: 10.1371/journal.pone.0066848. eCollection 2013. PMID 23990869